CLINICAL TRIAL: NCT06746831
Title: The Low-Down on Methamphetamine Isomers: Prevalence and Pharmacology in Humans
Brief Title: Methamphetamine Isomer Pharmacology in Humans
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: U.S. Department of Justice (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2024-1164; Protocol Version 2/12/25 (Other: UW Madison); A523000 (Other: UW Madison)
Record Dates: First submitted 2024-12-09; First posted 2024-12-24 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Methamphetamine
Keywords: pharmacology; meth; isomers

STUDY DESIGN:
Intervention Model Description: Double-blind crossover study design.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- S-Meth, R-Meth, Racemic Isomer (Experimental): First visit: Administer S-Meth, then at least 7 days later Second visit: Administer R-Meth, then at least 7 days later Third visit: Administer (1:1) racemic methamphetamine
  Interventions: Drug: S-(+)-methamphetamine; Drug: R-(-)-methamphetamine; Drug: 1:1 racemic mixture of two isomers
- R-Meth, Racemic Isomer, S-Meth (Experimental): First visit: Administer R-Meth, then at least 7 days later Second visit: Administer (1:1) racemic methamphetamine, then at least 7 days later Third visit: Administer S-Meth
  Interventions: Drug: S-(+)-methamphetamine; Drug: R-(-)-methamphetamine; Drug: 1:1 racemic mixture of two isomers
- Racemic Isomer, S-Meth, R-Meth (Experimental): First visit: Administer (1:1) racemic methamphetamine, then at least 7 days later Second visit: Administer S-Meth, then at least 7 days later Third visit: Administer R-Meth
  Interventions: Drug: S-(+)-methamphetamine; Drug: R-(-)-methamphetamine; Drug: 1:1 racemic mixture of two isomers

INTERVENTIONS:
Drug: S-(+)-methamphetamine — 15 mg
  Other Names: S-Meth
Drug: R-(-)-methamphetamine — 15 mg
  Other Names: R-Meth
Drug: 1:1 racemic mixture of two isomers — 15 mg R-Meth + 15 mg S-Meth

SUMMARY:
This study is being done to understand the metabolism and impairment profile of methamphetamine (meth). Meth exists as two chemical structures that are mirror images of each other: R-meth and S-meth. S-meth is a strong central nervous system stimulant and used to treat attention deficit disorder (ADD). R-meth is not a strong central nervous system stimulant and is available over-the-counter in nasal decongestant sprays.17 healthy participants will be enrolled for 3 study visits and on study for up to 12 weeks.

DETAILED DESCRIPTION:
Double-blind crossover study design. Healthy volunteers will attend three study drug administration visits, at least 7 days apart, in which methamphetamine isomer pharmacology will be assessed following intravenous administration of (1) S-(+)-methamphetamine, (2) R(-)-methamphetamine, or (3) a (1:1) racemic mixture of R-(-)- and S-(+)-methamphetamine. The order of these interventions will be counterbalanced across participants. Serial blood samples will be drawn during each dosing visit and compared with concurrent dried blood spots from a finger stick, oral fluid collections, and pooled urine specimens.

Primary Objective

* Characterize the pharmacokinetics of acute S-(+)-methamphetamine administration.
* Characterize the pharmacokinetics of acute R-(-)-methamphetamine administration.
* Characterize the pharmacokinetics of acute racemic (1:1) R-(-)- and S-(+)-methamphetamine administration.

Secondary Objectives

* Assess for evidence of stereo-selective metabolic pathways.
* Assess for evidence of subjective, cognitive, or physiological effects from acute R-(-)-methamphetamine administration.
* Assess for evidence of more than additive effects when administering racemic methamphetamine.

Correlative Objectives

* Compare biological methamphetamine and metabolite concentrations in surveyed biological matrices (i.e., plasma, whole blood, oral fluid, dried capillary blood spots, and urine) over time.
* Compare cognitive and subjective effects of acute S-(+)-methamphetamine, R-(-)-methamphetamine, and racemic methamphetamine administration.

ELIGIBILITY:
Inclusion Criteria:

* Good mental health as determined by self-reported responses to the Psychopathology Screener
* Absence of any major cardiac, neurologic, psychiatric, oncologic, endocrine, metabolic, renal, or hepatic disease as determined by self-reported responses to the Medical History Screener
* English-speaking (able to provide consent and complete questionnaires)
* Written Informed Consent

Exclusion Criteria:

* Any serious prior adverse response to sympathomimetic agents or amphetamine analogs
* History of or current substance use disorder as determined by self-reported responses to the Internalizing, Externalizing, and Substance Use Disorder Screener
* Pregnancy or lactation (pregnancy test, if needed)
* Use of medications that may impact cognition or metabolism (e.g., mood stabilizers, sedatives)
* Dependent on prohibited concomitant therapy that cannot be withheld for 48 hours prior to and during study visits.

Ages: 21 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | pre-dose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48 hours
  The pharmacokinetic analysis relies on observed drug and metabolite concentration measurements over time and across biological matrices (plasma, whole blood, dried capillary spots, oral fluid, urine) included in this study.
Area under the concentration versus time curve (AUC) | pre-dose, 0, 0.5, 1, 1.5, 2, 3, 4, 5, 6, 8, 10, 12, 16, 20, 24, 30, 36, 42, 48 hours
  The pharmacokinetic analysis relies on observed drug and metabolite concentration measurements over time and across biological matrices (plasma, whole blood, dried capillary spots, oral fluid, urine) included in this study.

SECONDARY OUTCOMES:
Cognitive Effects: Divided Attention Task (DAT) | Visit 1 (baseline), Visit 2 (week 1), Visit 3 (week 2)
  The DAT requires participants track a moving stimulus on a computer screen while simultaneously monitoring numbers located in the corners of the screen. Participants must respond to target numbers as they appear, and the task quantifies mean distance of the mouse cursor from the center of the target stimulus.
Cognitive Effects: Digital Symbol Substitution Task (DSST) | Visit 1 (baseline), Visit 2 (week 1), Visit 3 (week 2)
  The DSST asks participants to recreate patterns of various shapes presented on a computer screen using the keyboard. The total number of correct patterns are recorded within 90 seconds.
Cognitive Effects: Paced Serial Addition Task (PASAT) | Visit 1 (baseline), Visit 2 (week 1), Visit 3 (week 2)
  The PASAT has participants view a string of single-digit numbers and calculate the sum of the two most recently presented numbers. The total number of correct trials out of 90 will be recorded.
Subjective Effects: Drug Effect Questionnaire (DEQ) | Visit 1 (baseline), Visit 2 (week 1), Visit 3 (week 2)
  Subjective current general effects will be measured by asking the participant to rate if they feel the drug effect, if they like/dislike the drug effect, if they feel high, and if they would like more of the drug. Effects will be measured on a scale from "not at all" anchored at 0 to "extremely" at 100.
Subjective Effects: Number of Participants Who Answer 'True' for Amphetamine-specific questions | Visit 1 (baseline), Visit 2 (week 1), Visit 3 (week 2)
  Participants will be asked 11 amphetamine-specific questions including feelings of pleasantness, excitability, memory, emptiness, body tingling, weird feeling, patience, and mental sharpness. Results are measured as either "true" (experiencing the specific state) or "false" (not experiencing the specific state). Number of participants who answered 'True' is reported here

CONTACTS AND LOCATIONS:
Overall Officials: Heather K Barkholtz, PhD, Principal Investigator — University of Wisconsin, Madison; David Leinweber, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No